CLINICAL TRIAL: NCT05576168
Title: Shanghai Tenth People's Hospital,School of Medicine,Tongji University
Brief Title: Related Mechanisms of RBP4 in Glycolipid Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Manna, Director, Shanghai 10th People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RBP4
Record Dates: First submitted 2022-09-28; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Beta Cell Dysfunction
Keywords: Retinol binding protein 4; beta cell dysfunction; glycolipid metabolism

STUDY DESIGN:
Intervention Model Description: Serum RBP4 level in patients with or without type 2 diabetes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T2DM group (Experimental): patients with T2DM
  Interventions: Biological: overexpression STRA6/miRNA3
- control group (Active Comparator): patients without T2DM
  Interventions: Biological: overexpression STRA6/miRNA3

INTERVENTIONS:
Biological: overexpression STRA6/miRNA3 — RBP4 express in patients with T2DM or not
  Other Names: RBP4 express in T2DM patients

SUMMARY:
Retinol binding protein 4 ( RBP4 ) is a newly discovered adipokine secreted by adipose tissue, which leads to insulin resistance ( IR ) and participates in the occurrence of T2DM. At present, it's not clear whether RBP4 can cause islet β cell dysfunction. The purpose of this study is to explore the role of serum apo-RBP4 in the pathogenesis of newly diagnosed T2DM patients.

DETAILED DESCRIPTION:
In recent years, with the improvement of living standards and lifestyle changes, the incidence of type II diabetes is increasing, and T2DM has become a worldwide disease that seriously endangers people ' s health. When patients with diabetes in the middle and late, the condition is often irreversible, and early if effective treatment, help to improve the condition in a timely manner, delay the development of the disease process. Therefore, early diagnosis and treatment is the key to prevention and treatment of diabetes. Years of studies have shown that insulin resistance and β-cell dysfunction are the two major mechanisms of type II diabetes. Previous studies on the pathogenesis of type II diabetes mostly focused on insulin resistance, and there are few studies on β-cell dysfunction. Therefore, the study of islet β-cell dysfunction is extremely important. According to previous studies, the investigator found that although insulin resistance exists in type II diabetes, also exists to the same extent in many people who do not have diabetes. These people may have or do not have metabolic syndrome. Therefore, insulin resistance alone cannot be the decisive pathogenic factor of type II diabetes, and the increasing facts indicate that the abnormality of islet cells, especially islet β cells, may be the central link in the pathogenesis of type II diabetes. Obviously, insulin resistance is the initiating factor of type II diabetes, and the normal function of islet β cells is the determinant of whether type II diabetes occurs : the occurrence of insulin resistance initiates the pathogenesis of type II diabetes, but if the islet β cells can maintain its compensatory ability, type II diabetes will not occur. Once its compensatory ability decreases, type II diabetes gradually occurs. Therefore, islet β cell dysfunction is the key to the pathogenesis of type II diabetes. Exploring the harmful factors that impair β-cell function is critical for early prevention and treatment of diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Prior to conducting any trial-related activities, including those conducted to assess the subject's eligibility Informed consent of the subject;
2. Aged 18-60 years at the time of screening;
3. The diagnosis of diabetes was defined as fasting blood glucose above 7.0mmol/ L twice on different days on a normal diet

Exclusion Criteria:

1. HIV, hepatitis B or C ( self-reported ) or active pulmonary tuberculosis history :
2. history of malignant tumor ;
3. Severe liver dysfunction or kidney disease ( AST or ALT > 3 times the normal upper limit, or eGFR < 30ml min 1.73 m2 ) ;
4. History of severe cardiovascular and cerebrovascular diseases ( angina pectoris, myocardial infarction or stroke ) in the past 6 months :
5. history of severe gastrointestinal disease or gastrointestinal surgery in the past 12 months ;
6. There are other diseases that affect glucose and lipid metabolism : hyperthyroidism, hypothyroidism, cortex Hyperalcoholism, etc. ;
7. Secondary diseases or drugs lead to obesity, including : elevated cortisol ( such as Cushing 's syndrome ), sagging Obesity caused by body and hypothalamus injury, obesity caused by weight loss drug reduction / discontinuation, etc.
8. Drugs affecting body weight or energy intake / energy expenditure were used within 3 months before screening, including :

Sex steroids ( intravenous, oral or intra-articular ), tricyclic antidepressants, for psychiatric disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
RBP4 | 3 years
  Retinol binding protein 4

SECONDARY OUTCOMES:
BMI | 3 years
  BMI=weight(kg)/heihgt(m)^2
TT | 3 years
  total testosterone in mmol/L
FBG | 3 years
  fasting blood-glucose in mmol/L
PBG | 3 years
  postprandial blood-glucose in mmol-L
FINS | 3 years
  fasting serum insulin in mU/L
PINS | 3 years
  postprandial serum insulin in mU/L
ALT | 3 years
  alanine aminotransferase in U/L
AST | 3 years
  aspartate aminotransferase in U/L
UA | 3 years
  Uric acid in umol/L
HOMA-IR | 3 years
  Homeostatic model assessment insulin resistance index=FBG*FINS/22.5
HbA1c(%) | 3 years
  Glycated hemoglobin
FT | 3 years
  free testosterone (nmol/L)
LDL-C | 3 years
  low-density lipoprotein cholesterol in mmol/L
HDL-C | 3 years
  Hight-density lipoprotein cholesterol in mmol/L
FSH | 3 years
  follicle-stimulating hormone in IU/L
TC | 3 years
  Total Cholesterol(mmol/L)
TG | 3 years
  Triglyceride(mmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Shen Qu, Dr, Study Chair — Department of Endocrinology,Shang hai Tenth People's Hostipal,Shang hai,Shanghai,China,200070
Locations (1):
- Xiaoyun Cheng, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Weng Q, Zhao M, Zheng J, Yang L, Xu Z, Zhang Z, Wang J, Wang J, Yang B, Richard Lu Q, Ying M, He Q. STAT3 dictates beta-cell apoptosis by modulating PTEN in streptozocin-induced hyperglycemia. Cell Death Differ. 2020 Jan;27(1):130-145. doi: 10.1038/s41418-019-0344-3. Epub 2019 May 16. PMID 31097787